CLINICAL TRIAL: NCT01428791
Title: BRIGHTEN Heart: Reducing Disparities in Late Life Depression and Metabolic Syndrome
Brief Title: Reducing Disparities in Late Life Depression and Metabolic Syndrome
Acronym: BRIGHTEN-Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1P50HL105189-01 (NIH)
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Depressive Symptoms; Metabolic Syndrome X; Overweight; Obesity; Hypertension; Hyperglycemia; Dyslipidemias
Keywords: Geriatrics; Older adults; Health Disparities; Health Services for the Aged; Interdisciplinary Health Team; Depressive symptoms; Metabolic Syndrome X; Overweight; Obesity; Hypertension; Hyperglycemia; Dyslipidemias
MeSH Terms: conditions — Depression; Metabolic Syndrome; Overweight; Obesity; Hypertension; Hyperglycemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generations older adult member program (Active Comparator): Rush Generations is a membership program for older adults, providing chronic disease prevention and management through educational programming, civic engagement, and individual and family consultations with social work staff.
  Interventions: Behavioral: Generations older adult membership program
- BRIGHTEN Heart Virtual Team (Experimental): BRIGHTEN Heart provides older adults with an interdisciplinary team evaluation of physical and mental health and on-going support for mental health and health behavior change for a minimum of six months. The five core components of the BRIGHTEN intervention consist of: 1) Assessment; 2) Virtual team case review; 3) Patient centered action planning; 4) Plan implementation, and; 5) When indicated, short-term evidence-based geriatric specialty psychotherapy.
  Interventions: Behavioral: BRIGHTEN Heart Virtual Team intervention

INTERVENTIONS:
Behavioral: Generations older adult membership program — Rush Generations is a membership program for older adults emphasizing chronic disease prevention and management through a wide range of health and aging-related programs. Participants assigned to the Generations intervention are actively encouraged to participate in activities, including:
  • RUSH-based lectures by experts in the fields of health and aging providing practical information and resources on physical and mental health, functional status, and social support. • Individual and family consultations with social work staff. • Health fairs with a variety of assessment services and information about community-based social service and health agencies. • Assistance with referral to community programs such as physical activity, driver safety events, and mind-body connection workshops.
  Arms: Generations older adult member program
Behavioral: BRIGHTEN Heart Virtual Team intervention — BRIGHTEN Heart provides an interdisciplinary team evaluation of physical and mental health and on-going support for mental health & health behavior change for 6 - 12 months, including:
  • Comprehensive health risk assessment by a licensed social worker, including physical, mental, and functional status. • Virtual team case review and recommendations by interdisciplinary team including psychologist, social worker, occupational therapist, pharmacist, chaplain, dietitian, geriatric psychiatrist, and patient's primary care physician. • Development of Patient Centered Action Plan, in which the social worker assists the patient in prioritizing recommendations. • Monthly telephone calls by the social worker to support implementation of Action Plan and Case Management. • Evidence Based Psychotherapy, as needed, delivered by supervised geriatric psychology and social work fellows.
  Arms: BRIGHTEN Heart Virtual Team

SUMMARY:
Linkages between depression and cardiovascular disease have been well documented. These appear to be more than associations, and may reflect causal relationships through a number of proposed pathways, including decreased physical activity, poor dietary habits, medication non-adherence, and a direct impact on inflammatory mediators. Older adults are affected by both depression and heart disease, with increased risk in African American and Latino elderly.

The BRIGHTEN-Heart trial tests the hypothesis that an enhanced primary care delivery system intervention which provides evidence-based, patient-centered mental health services targeting depression and cardiovascular risk factors can reduce the risk of development of cardiovascular disease in low-income elderly blacks and Hispanics. BRIGHTEN stands for Bridging Resources of a Geriatric Health Team via Electronic Networking, and in this intervention, specialty providers including geropsychologists, social workers, pharmacists, nutritionists, chaplains, occupational therapists, and others collaborate via the internet as a virtual team. The study will determine if such a virtual interdisciplinary clinical team collaboration can reduce depression in older (age ≥ 65) minority adults with comorbid depression and metabolic syndrome.

DETAILED DESCRIPTION:
Chicago has been characterized as one of America's most segregated cities, with many neighborhoods characterized by black and Hispanic populations living in concentrated pockets of poverty. In addition to lowered socioeconomic status, these neighborhoods are also characterized by remarkable health disparities relative to wealthier, predominantly white neighborhoods only a few miles away. Disparities in access to health services contribute to these poorer health outcomes, but are not wholly explanatory.

For cardiovascular disease, the leading cause of death in the US, both black and Hispanic adults have elevated rates of many major risk factors including physical inactivity, obesity, elevated levels of Fasting Blood Glucose, and dyslipidemia. Blacks also have elevated rates of hypertension, and experience well-documented excess mortality rates. Experts are anticipating that, given high prevalence of risk factors, most importantly the metabolic syndrome, similar disparities in cardiovascular mortality may soon emerge for Hispanics as well.

Beyond cardiovascular disease, these populations face psychosocial challenges such as poverty, unemployment, societal racism, and high rates of major and traumatic life stress, all of which can contribute to high rates of depression and anxiety symptoms. Even the physical environment adds to the levels of stress: empty buildings that can become criminal and drug havens, boarded up storefronts, lack of groceries providing access to fresh fruits and vegetables (so-called "food deserts"). Disparities in access to health services, and these environmental conditions, as well as personal and familial factors associated with poverty are related to health disparity outcomes in complex ways that are only beginning to be understood.

Linkages between depression and cardiovascular disease have been well documented. These appear to be more than associations, but may reflect causal relationships through a number of proposed pathways, including decreased physical activity, poor dietary habits, medication non-adherence, and a direct impact on inflammatory mediators.

Aging is often associated with worsening of health disparities. The most vulnerable subpopulation among the urban poor are the elderly, as they are naturally vulnerable due to old age, compounded by lifetime exposure to poverty, and diminished defenses against violence in their homes or neighborhoods, including routes to health service providers.

To date, health care interventions targeting specific individual risk factors in the elderly have had only limited success in reducing health disparities in cardiovascular disease. The investigators hypothesize that this is due to two reasons. First, changes in the healthcare system are needed that feature multidisciplinary teams rather than individual practitioners. Second, treatment of cardiovascular risk factors requires attention to the patient's emotional state to guard against the possibility that providers and patients are working at cross-purposes; that is, the provider wants the patient to take action to improve long-term survival, while the patient is experiencing low self-esteem, hopelessness, helplessness, or even a passive or active wish to die. Reducing the risk of heart disease in this complex bio-psychosocial context requires more than prescribing the right medication or recommending that individuals modify their diet and exercise. The investigators hypothesize that a multi-level intervention targeting both the healthcare system and the individual's psychosocial and behavioral risk factors may succeed where past interventions have failed.

The investigators therefore propose testing the hypothesis that an enhanced primary care delivery system intervention which provides evidence-based, patient-centered mental health services targeting depression and cardiovascular risk factors can reduce the risk of development of cardiovascular disease in low-income elderly blacks and Hispanics. Researchers at Rush University Medical Center have developed and tested several "virtual" interdisciplinary team interventions, in which healthcare providers communicate as a team via e-mail, telephone, fax, or video conferencing. The first of these, the Virtual Integrated Practice project demonstrated that primary care practices could partner with community-based teams to improve care of older adults with chronic illness. A subsequent program called BRIGHTEN (Bridging Resources of a Geriatric Health Team via Electronic Networking) enhanced the assessment and treatment of late life depression and anxiety in primary care. The proposed "BRIGHTEN Heart study" will determine if a virtual interdisciplinary clinical team (BRIGHTEN Heart) can reduce depression in older (age ≥ 65) minority adults with comorbid depression and metabolic syndrome. The overall purpose of this study is to reduce racial disparities in cardiovascular morbidity and mortality in black and Hispanic elderly by effectively controlling behavioral and psychosocial risk factors.

A second, exploratory purpose of the study is to better understand the impact of current major stressors and lifetime and current traumatic stressors, as these may be "hidden" factors that impact emotional state, individual behavior, access to care, and intervention adherence. It is our goal to them incorporate what the investigators learn about the impact of major and traumatic stressors into later intervention as part of our overall Center efforts.

Study Hypothesis:

Compared to an educational group, older minority patients with symptoms of depression and comorbid metabolic syndrome receiving the BRIGHTEN Heart virtual team intervention will demonstrate

1. Significant reductions in symptoms of depression [Primary trial outcome]
2. Significant reductions in metabolic syndrome
3. Improved adherence with medications prescribed for medical illnesses

Primary Aim

1. To determine whether BRIGHTEN Heart can reduce depression symptoms in older adults with the metabolic syndrome

   Secondary Aims
2. To determine whether the BRIGHTEN Heart intervention can result in reduced prevalence of metabolic syndrome as compared to a control population
3. To test the mediating hypothesis that the BRIGHTEN Heart intervention results in improvements in adherence with medications

   Exploratory Aim
4. To explore the impact of trauma and major life stressors on the results of the intervention

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years of age.
* Overweight or Obese as documented by BMI greater than 25.0.
* Presence of Depression symptoms, as determined by having a PHQ-9 score of 8 or more.
* Receiving primary care through a participating safety net clinic (public clinic or FQHC)

Exclusion Criteria:

* Below the age of 60 years old at time of enrollment.
* Lack decisional capacity (due to dementia, active psychosis, or other cause).
* Are currently under active behavioral treatment of a psychologist or psychiatrist for any reason.
* Lack regular access to a telephone in their home (including cell phone).
* Are enrolled in another intervention trial

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06-30 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Clinical Depression Scores, as measured by PHQ-9 | 6 months
  Depression has been shown to double both the risk of developing heart disease and mortality risk for persons who do develop heart disease. The Primary Aim of the trial is to document reduction in symptoms of depression in persons receiving the intervention, relative to the control group. The PHQ-9 instrument is the most widely used symptom measure of depression, and has been validated across multiple populations, and in a Spanish-translation as well

SECONDARY OUTCOMES:
Cardiometabolic risk factors | 6 months
  Risk for the development of heart disease will be compared via clinical measures and blood tests. Clinical measurements include Blood Pressure, Weight, and Waist Circumference. Blood tests include Hemoglobin A1c, HDL Cholesterol, LDL Cholesterol, and hsCRP.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Rothschild, MD, Principal Investigator — Department of Preventive Medicine, Rush University Medical Center; Erin Emery, PhD, Principal Investigator — Department of Behavioral Sciences, Rush University Medical Center
Locations (2):
- United States (2):
  - Cook County Health and Hospital System, Chicago, Illinois
  - Mercy Hospital and Health System, Chicago, Illinois

REFERENCES:
- [Derived] Emery-Tiburcio EE, Rothschild SK, Avery EF, Wang Y, Mack L, Golden RL, Holmgreen L, Hobfoll S, Richardson D, Powell LH. BRIGHTEN Heart intervention for depression in minority older adults: Randomized controlled trial. Health Psychol. 2019 Jan;38(1):1-11. doi: 10.1037/hea0000684. Epub 2018 Nov 1. PMID 30382712